CLINICAL TRIAL: NCT02992834
Title: Anti-CD19:TCRζ Chimeric Antigen Receptor-T Cells in the Treatment for Chemotherapy-resistant or Refractory CD19+B Cell Lymphoma:a Double-arm, Single Center, Open-label Clinical Trial
Brief Title: Anti-CD19:TCRζ Chimeric Antigen Receptor-T Cells in the Treatment for CD19+ B Cell Lymphoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: jiangjingting (Other)
Responsible Party: Sponsor-Investigator, jiangjingting, Professor, The First People's Hospital of Changzhou
Organization: The First People's Hospital of Changzhou (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAA
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Lymphoma, B Cell
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IL-2 pre-treated CD19 cells (Active Comparator): Initial therapy: IL-2 (interleukin,IL)stimulated, CD28-ζ-vector (cluster of differentiation 28,CD28)transfected T cells(TCRζ chimeric antigen receptor-T cell)， were administered at 1×106/kg by single infusion
  Interventions: Biological: IL-2 pre-treated CD19 cells
- IL-7/IL-15 pre-treated CD19 cells (Active Comparator): Initial therapy: IL-7/IL-15 stimulated, CD28-ζ-vector transfected T cells(TCRζ chimeric antigen receptor-T cell)， were administered at 1×106/kg by single infusion
  Interventions: Biological: IL-7/IL-15 pre-treated CD19 cells

INTERVENTIONS:
Biological: IL-2 pre-treated CD19 cells — IL-2 stimulated, CD28-ζ-vector transfected T cells(TCRζ chimeric antigen receptor-T cell)， were administered at 1×106/kg by single infusion
  Arms: IL-2 pre-treated CD19 cells
Biological: IL-7/IL-15 pre-treated CD19 cells — IL-7/IL-15 stimulated, CD28-ζ-vector transfected T cells(TCRζ chimeric antigen receptor-T cell)， were administered at 1×106/kg by single infusion
  Arms: IL-7/IL-15 pre-treated CD19 cells

SUMMARY:
This study aims to evaluate the safety, efficacy and duration of response of CD19 Chimeric Antigen Receptor (CAR) redirected allogeneic T-cells in patients with chemotherapy-resistant or refractory CD19+ B cell lymphoma.

DETAILED DESCRIPTION:
This is a single-centre, randomised, open label Phase I clinical trial of CD19 Chimeric Antigen Receptor (CAR) T-cells (CD19 CAR T-cells) in patients with chemotherapy-resistant or refractory CD19+ B cell lymphoma. Following informed consent and registration to the trial, Patients will receive the allogeneic CD19 CAR T-cells following lymphodepleting chemotherapy. The study will evaluate the safety, efficacy and duration of response of the CD19 CAR T-cells in patients with chemotherapy-resistant or refractory CD19+ B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Enrollment for enough male or female patients with CD19+ hematological malignancies, without regimens for cure (autologous or allogeneic stem cell transplantation), and having a poor prognosis (several months to 2 years) under current optional regimens

1. Age ranges from 18 to 70 years old
2. Expected survival time longer than 12 weeks
3. Performance status score 0-2
4. Pathologically confirmed CD19+ lymphoma (CD19+ follicular lymphoma, Mantle cell lymphoma, diffuse large B cell lymphoma) and meets at least one of follows:

   1. having received at least 2-4 cycles of combined chemotherapy (excluding monoclonal antibody monotherapy, such as rituximab) but do not reach a complete response; recurrent disease; not applicable for conventional stem cell transplantation; being partial responsible or stable but not complete responsible after the latest therapy
   2. recurrence develops after stem cell transplantation
   3. diagnosis confirmed but refusing to receive conventional therapy
5. Creatinine<2.5 mg/dl；
6. alanine aminotransferase/aspartate aminotransferase lower than 3 folds of normal range
7. Bilirubin<2.0 mg/dl；
8. Venous channel available and no contraindications for leukocyte collection
9. Reliable contraception from the beginning to 30 days after discontinuation of therapy
10. Informed consent signed

Exclusion Criteria:

1. Central nerve system invasion with symptoms
2. Other concurrent uncontrolled malignancies
3. Hepatitis B infection or active period of hepatitis C, HIV infection
4. Other uncontrolled diseases hampering the intervention in the study
5. Coronary heart disease, angina, myocardial infarction, arrhythmia, cerebral thrombosis, cerebral hemorrhage and other serious cardiovascular or cerebrovascular diseases.
6. Grade 2-3 or uncontrolled hypertension
7. History of uncontrolled mental disease
8. Not suitable for participation judged by researchers
9. Immunosuppressive agents administered due to organ transplantation, not including recent or current inhaled corticosteroid
10. Medical history of mental diseases or abnormities of lab tests might increase the risks of participation in study or drug administration, or interfering the results
11. Screening suggesting transfection efficiency of targeting cells lower than 30% or cell expansion deficiency under CD3/CD28 (cluster of differentiation 3,CD3)stimulation (less than 5 folds)
12. Unstable pulmonary embolism, deep venous thromboembolism or other major arterial/venous thromboembolism events develop in 30 days before the randomization. If anti-coagulation therapy is received, the treatment dose should reach stability before the randomization.
13. Pregnancy or lactation, or pregnancy planned during the study or in 2 months after the study
14. Reliable contraception not accepted during the study or in 2 months after the study. Female subjects are required to provide negative results from serum or urine pregnancy test 48 hours before therapy
15. Systematic active or uncontrolled infection (excluding infection of urinary tract or upper respiratory tract infection) in 14 days before the randomization
16. Informed consent not signed or study rules violated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-12; Primary Completion 2020-08 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 year

SECONDARY OUTCOMES:
progression-free survival | 56 day
Objective Response Rate | 56 day

CONTACTS AND LOCATIONS:
Overall Officials: Jingting Jiang, Professor, Principal Investigator — The First People's Hospital of Changzhou
Locations (1):
- First People's Hospital of Changzhou, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rafiq S, Purdon TJ, Daniyan AF, Koneru M, Dao T, Liu C, Scheinberg DA, Brentjens RJ. Optimized T-cell receptor-mimic chimeric antigen receptor T cells directed toward the intracellular Wilms Tumor 1 antigen. Leukemia. 2017 Aug;31(8):1788-1797. doi: 10.1038/leu.2016.373. Epub 2016 Dec 7. PMID 27924074
- [Background] Minagawa K, Jamil MO, Al-Obaidi M, Pereboeva L, Salzman D, Erba HP, Lamb LS, Bhatia R, Mineishi S, Di Stasi A. In Vitro Pre-Clinical Validation of Suicide Gene Modified Anti-CD33 Redirected Chimeric Antigen Receptor T-Cells for Acute Myeloid Leukemia. PLoS One. 2016 Dec 1;11(12):e0166891. doi: 10.1371/journal.pone.0166891. eCollection 2016. PMID 27907031